CLINICAL TRIAL: NCT04679649
Title: Physiotherapy of Axial Spondyloarthritis - PaxSpA Trial A: Manual Spinal Mobilisation in Patients With Axial Spondyloarthritis
Brief Title: Physiotherapy of Axial Spondyloarthritis
Acronym: PaxSpA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal United Hospitals Bath NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PaxSpA V5 28072020
Record Dates: First submitted 2020-11-16; First posted 2020-12-22 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Axial Spondyloarthritis
Keywords: physiotherapy; manual mobilisation; axial spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Intervention Model Description: Pragmatic randomised controlled clinical trial (RCT) with secondary element of observational cohort trial in line with the "Trials within Cohort design" (TwiCs). Trial A is Manual mobilisation of the spine.
Who Masked: Participant, Outcomes Assessor
Masking Description: Batch randomisation - computer generated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial A - Intervention Group (manual mobilisation) (Experimental): Participants will continue to receive routine care and 13 sessions of manual spinal mobilisation will be administered over a 6 months period to compare routine care vs routine care plus manual spine mobilisation physiotherapy.
  Interventions: Other: Manual spinal mobilisation physiotherapy
- Trial A - Control Group (routine care) (No Intervention): Participants in control group will continue to receive routine care, and routine care measurements for axial spondyloarthritis will be taken at baseline, 3 months and 6 months plus follow up.

INTERVENTIONS:
Other: Manual spinal mobilisation physiotherapy — Manual spinal mobilisation is a physiotherapy technique to improve spinal mobility by gently applying pressure manually on the each segmental vertebrae by hands-on treatment of a physiotherapist.
  Other Names: "Maitland's" mobilisations
  Arms: Trial A - Intervention Group (manual mobilisation)

SUMMARY:
This protocol is for a pragmatic randomised controlled clinical trial (RCT) with a manual spinal mobilisation (MSM) intervention for patients with axial spondyloarthritis (axSpA), embedded in a Trials within Cohort (TwiCs) design. This trial might appear as a standardised RCT but there is a secondary element - an observational cohort the trial is embedded in. Trial A is the first (of possibly several) embedded pragmatic RCTs involving physiotherapy interventions that may identify therapies that will help improve outcomes for patients with axSpA.

The investigators are seeking to improve outcomes for these patients by comparing different physiotherapy interventions in subsequent trials with standard of care (SoC) physiotherapy. Trial A will compare routine care vs routine care plus MSM physiotherapy attempting to answer the primary research question if MSM on patients with axSpA improves spinal mobility.

In order to recruit patients and obtain outcomes for Trial A (n=70), the investigators will first recruit up to 300 axSpA patients receiving care at the Royal National Hospital for Rheumatic Diseases (RNHRD) in Bath into a cohort and observe their standard of care outcomes. This will allow to answer the cohort's research question of "How does SoC physiotherapy in patients with axSpA reflect in data collected routinely on outcomes of the disease?" Patients will be asked to consent to provide routine observational data on their wellbeing, be approached to take part in future trials of interventions which aim to improve outcomes for patients with axSpA, and not be approached unless they are offered the physiotherapy trial intervention. This highly pragmatic method of providing information and seeking consent replicates the informed consent procedures in routine care clinical settings. This study is aimed to last three years, with individual trials of 40-70 participants, ranging between three to six months duration of therapy intervention in addition to routine care.

DETAILED DESCRIPTION:
A single pragmatic randomised controlled clinical trial (RCT) (Trial A) which is embedded in a series of pragmatic trials within the Trials within Cohort (TwiCs) design of the PaxSpA study. This trial will compare manual spinal mobilisation (MSM) intervention for patients with axial spondyloarthritis (axSpA) to routine care alone.This trial might appear as a standardised RCT but there is a secondary element - an observational cohort the trial is embedded in. Trial A is the first (of possibly several) embedded pragmatic RCTs involving physiotherapy interventions that may identify therapies that will help improve outcomes for patients with axSpA. The cohort might seem as an unnecessary add-on to what could be conducted as a standalone standardised RCT, but it has a few important advantages. By having a cohort the investigators can observe routine care physiotherapy outcomes for a large cohort giving data from a large number of patients. That data can be used to compare to across a range of interventions, as each embedded trial will use the same outcome measures and therefore results are comparable across trials to give a broader view of the care of this chronic progressive condition - axial Spondyloarthritis. The other advantage for having for having the cohort is to be able to have a control group receiving standard of care without having disappointment bias for not being in the intervention arm, as physiotherapy interventions can be very difficult to blind participants. The investigators plan to establish an observational cohort of 300 patients with axial spondyloarthritis (axSpA) currently treated at the RUH NHS Trust in Bath and observe their outcomes over the duration of the study, as a cornerstone for our "Trials within cohort" (TwiCs) study PaxSpA. Cohort patients will be asked to consent to (i) provide observational data on their wellbeing (standard routine axSpA PROM), (ii) be approached to take part in future trials of interventions which aim to improve outcomes for patients axSpA, and (iii) not be approached unless they are offered an experimental (i.e. non routine) intervention. Post randomisation, only those randomly selected to an experimental (non-routine) intervention will informed about the experimental interventions and asked for their 'clinical' consent to receive these intervention (i.e. Trial A: manual mobilisation). This method is known as the Trials within Cohorts (TwiCs) method and is currently being used in over 70 studies worldwide, including many in the United Kingdom (UK) and Canada. This method of providing information and seeking consent replicates the informed consent procedures in routine care and has several benefits. Firstly, it avoids unnecessary expectation and disappointment regarding the experimental interventions. Secondly, clinicians do not have to spend time explaining interventions to patients who will not be offered the intervention post randomisation. Thirdly, it enables fast and efficient recruitment to both trials.

The investigators will then conduct the first of possibly several embedded pragmatic randomised controlled trials of adjunctive physiotherapy for patients with axSpA: Trial A will compare routine care vs routine care plus manual spinal mobilisation physiotherapy. The hypothesis for trial A assumes manual spinal mobilisation will improve function, decrease pain and decrease disease activity, but primarily increase spinal mobility, as shown in previous trials to be the case when specific parts of the spine received manual mobilisation.

The study design and methodology has been chosen because of its highly pragmatic character in a clinical setting of a chronic condition. Physiotherapy in axSpA consists of a variety of treatment options to research and outcomes for each intervention can be compared to the routinely taken outcome measures across the cohort to identify and compare benefits/challenges of different interventions. The TwiCs design has been shown to be particularly suitable for chronic conditions, where different treatments are provided to inform clinical practice, and therefore the investigators identified this design to be best suited to meet the aims and objectives our study (also see second paragraph above).

The justification for including control arms to a trial:

The control arm is important for comparison of outcomes and to increase the validity of our study. The control arm will receive standard of care as usual (as will the intervention group), without the additional intervention, therefore the difference in results between the groups will indicate the effect of the trial intervention, enabling to inform clinical practice. Additionally, it is very challenging to blind participants and researcher to physiotherapy interventions, so randomisation with a control group gives our study a sound methodology.

Randomisation will be achieved my random computer allocation in a staged (phased) randomisation process. Initially all cohort participants will get screened for eligibility for trial A and if successful, included into the eligible trial cohort. For trial A the investigators aim to recruit 12 participants per stage/batch into the manual mobilisation trial for six batches (up to 70 participants). For each batch, six participants will get randomly selected from the eligible trial cohort to be offered to receive the intervention. The remaining six participants that were not selected will function as controls. On average the investigators will aim to recruit a new batch every two weeks to start the initially more frequent intervention (from biweekly to monthly over six months) in stages. Therefore, all participants should have been randomised and started the trial within the first 3-4 months of the start of the trial. This phased randomisation/ recruitment to the trial is a due to limited resources and time restraints.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years of age from the RUH Bath National Health Service (NHS) Foundation Trust Rheumatology service based at RNHRD who fulfil the modified New York Criteria or the Assessment of SpondyloArthritis international Society (ASAS) axial spondyloarthritis criteria giving written consent for participation.

Exclusion Criteria:

* Mechanical spinal disease causing red flag symptoms such as cauda equina syndrome
* Age >70
* Pregnancy or breastfeeding
* Any malignancy
* Moderate coexistent other inflammatory conditions (such as rheumatoid arthritis, vasculitis or connective tissue disease, in order to minimise the effect particularly of inflammation). However clinical judgement might be used to judge the severity in some patients as to whether they are safe to be included in a trial.
* Any bridging syndesmophytes in the spine, to avoid the risk of causing vertebral fractures or instability

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change of Spinal Mobility | baseline, 6 months, and follow-up at 12 months
  Spinal mobility will be measured using inertial measurement unit sensors; Electro muscle stimulation (EMS) for muscle activity
Change of Spinal Mobility | baseline, 3 months & 6 months, and follow-up at 12 months
  Spinal mobility will be measured using the Bath Ankylosing Spondylitis Metrology Index (BASMI), scored on the mean of 5 items out of 0-10 (minimum value 0 maximum value 10), '0' being the best outcome and 10 being the worst outcome.

SECONDARY OUTCOMES:
Change of Disease Activity | baseline, 3 month, 6 month, 12 month
  Disease activity using BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) scored on the mean of 6 items out of 0-10 (minimum value 0, maximum value 10), '0' being the best outcome and 10 being the worst outcome.
Change of Functional limitation | baseline, 3 month, 6 month, 12 month
  Functional limitation is measured using BASFI (Bath Ankylosing Spondylitis Functional Index) scored on the mean of 10 items out of 0-10 (minimum value 0, maximum value 10), '0' being the best outcome and 10 being the worst outcome.
Change of Quality of Sleep (PROM) | baseline, 3 month, 6 month, 12 month
  measured using the Jenkins Sleep Evaluation Questionnaire (JSEQ) PROM The JSEQ is a 4-item self-report questionnaire designed to measure how often a subject has experienced sleep problems in the past month. JSEQ items evaluate trouble falling asleep, staying asleep, waking up several times, and awakening unrefreshed with each item scored on a 5-point Likert scale from 0 = "not at all" to 5 = "22-31 days." Scores vary from 0 to 20 with higher scores indicating more frequent sleep problems (worse outcome) and lower scores indicate a better outcome.
  '0' being the best outcome and 10 being the worst outcome.
Change of Quality of Life (PROM) | baseline, 3 month, 6 month, 12 month
  measured using the Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL). Each statement on the ASQoL is given a score of "1" or "0". A score of "1" is given where the item is affirmed, indicating adverse QoL. All item scores are summed to give a total score or index. Scores can range from 1 (good QoL outcome) to 18 (poor QoL outcome).
Change of Work Productivity (PROM) | baseline, 3 month, 6 month, 12 month
  measured using the Work Productivity and Activity Impairment Questionnaire (WPAI). WPAI scores are based on 1-item (presentism, activity impairment), 2-items (absenteeism) and multiple items (overall work productivity); a score cannot be calculated if there is a missing response to the corresponding item. The WPAI-GH consists of six questions: 1 = currently employed; 2 = hours missed due to health problems; 3 = hours missed other reasons; 4 = hours actually worked; 5 = degree health affected productivity while working (using a 0 to 10 Visual Analogue Scale (VAS)); 6 = degree health affected productivity in regular unpaid activities (VAS).scores are expressed in percentage (0-100) with a lower percentage indicating a better outcome and higher percentage indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Carter, Study Director — Royal United Hospitals Bath NHS FT
Locations (2):
- United Kingdom (2):
  - Sports Physiotherapy Calne, Calne, UK
  - Royal National Hospital for Rheumatic Diseases (RNHRD), Bath, Wiltshire

IPD SHARING:
Plan to Share IPD: Yes
Dr Sengupta has established a national and international panel of collaborators in the field of axial spondyloarthritis. We will therefore try to maintain our links with other experts in the field who are conducting cutting edge research in axSpA. Thus, the data collected as part of this study may be used in further research.
  Anonymised data may be shared with other researchers investigating non-pharmaceutical therapies in spondyloarthropathy.
  Requests for data would be evaluated on the basis of the research objectives of the intended project and any conflict of interests involved. If approved, recipients of data must forward copies of their protocol and ethics approval if appropriate to Dr Sengupta and the sponsor (RUH Bath NHS Foundation Trust Rheumatology service based at the RNHRD).
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Study Protocol and Consent form become available once recruitment has started. Clinical Study report becomes available on study conclusion.
Access Criteria: request access through Dr Raj Sengupta